CLINICAL TRIAL: NCT05308901
Title: A Phase II Clinical Trial Evaluating The Combination Of Lenvatinib Plus Pembrolizumab In Patients With Treatment Naive Metastatic Uveal Melanoma
Brief Title: Lenvatinib Plus Pembrolizumab In Patients With Immune Checkpoint Inhibitor Naïve Metastatic Uveal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021000802
Record Dates: First submitted 2022-01-11; First posted 2022-04-04 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Melanoma, Uveal
Keywords: Melanoma; Uveal; Pembrolizumab; Phase 2; Lenvatinib
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Lenvatinib (Experimental): Lenvatinib 20 mg daily plus pembrolizumab 200 mg IV every 3 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV every 3 weeks for a maximum of 2 years.
  Other Names: Keytruda
Drug: Lenvatinib — 20 mg daily for a maximum of 2 years.

SUMMARY:
The purpose of this study is to evaluate the efficacy of lenvatinib and pembrolizumab to treat metastatic uveal melanoma.

DETAILED DESCRIPTION:
This is a phase II, single arm, single institution clinical trial. Adults (age≥18 years-old) with immune checkpoint inhibitor naïve metastatic uveal melanoma will be evaluated for eligibility. Eligible participants will be treated with the combination of Lenvatinib 20 mg daily + pembrolizumab 200 mg IV every 3 weeks for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic uveal melanoma will be enrolled in this study.
* Male participants must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days after the last dose of Lenvatinib and refrain from donating sperm during this period.
* Female participants are eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
  2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days post pembrolizumab or post Lenvatinib whichever occurs last.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on iRECIST. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. If slides are only available, ten slides would be required. Newly obtained biopsies are preferred to archived tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Have adequate organ function as defined in the following table (Table 2). Specimens must be collected within 7 days prior to the start of study intervention.
* Subjects must agree to undergo paired fresh tumor biopsy specimens (to be collected pre-treatment and day #15). Subjects with tumor metastases that are not amenable to image guided biopsies or who have a contraindication to biopsy (including but not limited to anticoagulation therapy that cannot be interrupted for a biopsy) are still eligible for participation in the clinical trial without undergoing biopsies.

Exclusion Criteria:

* A WOCBP who has a positive serum pregnancy test within 24 hours prior to the first dose of study intervention (see Appendix 3).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137). Prior therapy with Tebentafusp is permitted. Prior liver directed therapy is permitted (including but not limited to radioembolization, chemoembolization, immunoembolization, radio-frequency ablation, external beam radiation and resection).
* Participants previously treated with radiation therapy must have recovered from all radiation-related toxicities and not require corticosteroids.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed-virus vaccines and mRNA vaccines are allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early stage bladder cancer, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* Uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
* Electrolyte abnormalities that have not been corrected
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
* Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
* Subjects having ≥2+ proteinuria on urine dipstick testing. However, subjects with ≥2+ proteinuria on urine dipstick testing may undergo a 24-hour urine collection for quantitative assessment of proteinuria. Subjects with <1 g/24-hour proteinuria are eligible for participation.
* Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy. Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]).
* Females of child-bearing potential must be willing to use effective contraception during study and for 120 days after the last dose
* The participant has severe hypersensitivity (≥Grade 3) to lenvatinib and/or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2027-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Taylor, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib
Started | 6
Completed | 0
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Population: Trial closed to enrollment early due to poor accrual.
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measure of functional status from scores ranging from 0 to 5. Baseline measure ECOG PS was collected during the screening physical exam.
  Participants
    ECOG PS 0 (Asymptomatic) | 6
    ECOG PS 1 (Symptomatic but completely ambulatory) | 0
    ECOG PS 2 (Symptomatic, <50% in bed during the day) | 0
    ECOG PS 3 (Symptomatic, >50% in bed, but not bedbound) | 0
    ECOG PS 4 (Bedbound) | 0
    ECOG PS 5 (Death) | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effect of Lenvatinib Plus Pembrolizumab on Progression Free Survival
Description: Progression free survival, defined as the time from enrollment to the first documented evidence of disease progression or death.
Time Frame: An average of 6 months and 7 days from the time of enrollment.
Measure: Mean (Full Range); unit: days
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 6
days | 165 [63 to 504]

2. Secondary Outcome: Evaluate the Objective Response Rate Resulting From Treatment With Lenvatinib Plus Pembrolizumab
Description: Objective response rate (complete and partial responses assessed by iRECIST)
Time Frame: 6 weeks after treatment discontinuation
Population: Tumor assessments were not completed for 2 patients after treatment discontinuation due to disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 4
Participants
  iCR (Complete Response) | 0
  iPR (Partial Response) | 0
  iSD (Stable Disease) | 3
  iUPD (Unconfirmed Progression) | 1
  iCPD (Confirmed Progression) | 0

3. Secondary Outcome: Evaluate the Effect of Treatment With Lenvatinib Plus Pembrolizumab on Overall Survival
Description: Overall survival, defined as the time from enrollment to death (resulting from any cause).
Time Frame: 12 weeks post treatment discontinuation
Measure: Mean (Full Range); unit: Days
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 6
Days | 287 [75 to 758]

4. Secondary Outcome: Evaluate the Safety and Tolerability of Treatment With Lenvatinib Plus Pembrolizumab in Patients With Metastatic Uveal Melanoma
Description: Number of participants who experienced dose reduction or treatment discontinuation due to treatment related adverse events (TRAE).
Time Frame: 30 days after last treatment dose, on average 5 months from the start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were collected during each visit and at end of treatment visit.
Arm/Group | Pembrolizumab + Lenvatinib
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic Hemorrhage (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=6)
Abdominal cramping (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (9)
Alanine aminotransferase increase (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
BUN increased (Investigations) | 1 (1)
Bursitis, L Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Callous (Skin and subcutaneous tissue disorders) | 1 (2)
Cold like symptoms (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dermatitis, rectum (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (6)
Displaced tooth (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Early satiety (Gastrointestinal disorders) | 1 (1)
Edema, limbs (General disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme, bilateral ankles (Skin and subcutaneous tissue disorders) | 1 (3)
Fatigue (General disorders) | 5 (10)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fracture, tooth (Injury, poisoning and procedural complications) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Gout, L big Toe (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2)
Immune mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Maculo-papular rash, left knee (Skin and subcutaneous tissue disorders) | 1 (1)
Mental fog (Psychiatric disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 5 (6)
Neoplasm, benign- Dentigerous cyst, R maxilla (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 3 (3)
Oral sensitivity (Gastrointestinal disorders) | 1 (1)
Pain of skin (tender/sensitive) (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Phytophotodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Pyuria (Renal and urinary disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Retinal ischemia (Eye disorders) | 1 (1)
Right Medial Meniscus Tear (Injury, poisoning and procedural complications) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tooth pain (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vasovagal Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (Investigations) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT05308901/Prot_SAP_000.pdf